CLINICAL TRIAL: NCT02034461
Title: Can an Array of Micro-electrodes Implanted in a Human Nerve Record Neural Signals and Provide Sensory Feedback Useful for Controlling a Prosthetic Device?
Brief Title: Micro-Electrodes Implanted in a Human Nerve
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This device feasibility study was using a microelectrode array device to determine
  viability of the product. Design and operating specification of the device were established. A new IDE
  trial has been initiated.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, M.D., University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 55621
Record Dates: First submitted 2013-05-03; First posted 2014-01-13 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Amputations; Peripheral Nerve Injury; Spinal Cord Injury
Keywords: Micro-Electrodes; Peripheral Nerve Injury; Amputation; Spinal Cord Injury
MeSH Terms: conditions — Peripheral Nerve Injuries; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acute surgical implantation (Experimental): The investigators will conduct three acute surgeries where a Utah slanted Electrode Array (USEA) will be implanted in volunteers who are about to undergo limb amputations. These acute implantations will provide the PI with human surgical experience in implanting USEAs and evaluating the containment system the investigators will be using to immobilize the implanted USEA in the nerve.
  Interventions: Device: Utah Slanted Electrode Array
- Implantation of a Utah Electrode Array (Experimental): The arm which has been amputated or has peripheral nerve trauma. Intervention include insertion of the Utah Slanted Electrode Arrays which will interact with nerve endings in order to gain knowledge about device feasibility and nerve stimulation.
  Interventions: Device: Utah Slanted Electrode Array

INTERVENTIONS:
Device: Utah Slanted Electrode Array — Microelectrode slanted arrays with a large number of electrodes will be surgically implanted into peripheral nerves of patients with limb amputations or peripheral nerve trauma.

SUMMARY:
The main objective of the intervention in the study is devise feasibility using high-count microelectrode arrays implanted into peripheral nerves of patients with limb amputations or peripheral nerve injury. These microelectrodes will be custom-made and are not available for commercial distribution. The investigators hypothesize that recording neural signals from a large number of microelectrodes will provide selective motor information in high enough numbers to allow control over future artificial devices with many moving parts, i.e. artificial limbs with shoulder, elbow, wrist, and/or individual fingers that move. These studies will also investigate to what extent microstimulation of nerve fibers can provide sensory feedback from a prosthetic limb.

The investigators will also conduct up to three acute surgeries where a Utah slanted Electrode Array (USEA) will be implanted in volunteers who are about to undergo limb amputations. These acute implantations will provide Dr. Hutchinson with human surgical experience in implanting USEAs and evaluating the containment system we will be using to immobilize the implanted USEA in the nerve.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age and less than 65 years of age
* amputations
* peripheral nerve injury
* twelve participants for the 30 day implantation/physiological experimentation study
* three participants for the acute surgical implantation part of the study

Exclusion Criteria:

* incarceration
* pregnancy
* inability to consent
* psychiatric comorbidity
* increase the risk of adverse effects of general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-04; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Device feasibility to collect data from peripheral nerves, and will consist of action potentials (mV) arising from the axons surrounding the tip of each electrode. | Up to 4 Week Follow-up
  Device feasibility evaluation to confirm design and operating specifications of the device to collect action potentials from peripheral nerves.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hutchinson, Principal Investigator — Orthopedic Surgery
Locations (1):
- The University Orthopaedic Center, Salt Lake City, Utah, United States